CLINICAL TRIAL: NCT05395039
Title: Communication in the Hospital: Impact on Patients With Alzheimer's Disease and Other Causes of Cognitive Impairments and Their Surrogate Decision Makers
Brief Title: Virtual Communication in the Hospital: Impact on Patients and Surrogates
Acronym: VCHIPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment effort yielded no enrollments, so this study was stopped. We are re-evaluating the study design.
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH); Indiana University Health (Other); Regenstrief Institute, Inc. (Other)
Responsible Party: Principal Investigator, Alexia M. Torke, Professor of Medicine, Associate Division Chief, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10893; K24AG053794 (NIH)
Record Dates: First submitted 2022-04-15; First posted 2022-05-27 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Communication; Anxiety; Depression; Distress, Emotional
MeSH Terms: conditions — Communication; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Intervention Group: VCHIPS Control Group: Usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care: Control Group (No Intervention): No interventions administered. Participant will receive usual care in the hospital.
- VCHIPS: Intervention Group (Experimental): Individuals in this group will work with a study nurse to schedule the intervention.
  Interventions: Other: VCHIPS

INTERVENTIONS:
Other: VCHIPS — Participants in this group will have the opportunity to receive virtual visits with the patient during the hospital stay, led by a study nurse.
  Arms: VCHIPS: Intervention Group

SUMMARY:
This is a pilot study of scheduled video/audio conferences by clinical navigators on the experience of surrogate decision makers for hospitalized older adults with Alzheimer's disease (AD), delirium, and other causes of cognitive impairment. The purpose of this study is to learn more about the experiences of surrogate decision makers of hospitalized older adults when they cannot be physically present with the patient in the hospital. We will conduct a randomized pilot study of virtual visits to connect the surrogate decision makers of incapacitated, hospitalized older adults with AD, delirium, and related causes of cognitive impairment with the patient and clinicians.

DETAILED DESCRIPTION:
As the COVID-19 pandemic exploded, hospitals across the globe completely excluded or severely limited family visitors. Thousands of patients have faced life-threatening illness or died without any loved ones at the bedside. Patients with AD were often unable to understand why their family members could not be present, leading to increased agitation. The calming presence that family often provide to hospitalized patients was missing. In addition to the tragedy for patients, family members were forced to address decisions about life-sustaining treatments without being able to see the patient or talk face to face with clinicians. As our knowledge of coronavirus transmission expanded, visitor restrictions have been relaxed in some cases but not eliminated. Urgent interventions are needed to mitigate the harm of these restrictions. While the future is uncertain, COVID-19 cases are rising across the country, suggesting that visitation will continue to be restricted. Additionally, our tertiary referral center often admits patients from across the state, limiting the ability of family members to be at the bedside. Harnessing virtual technologies has the potential to enhance surrogate/clinician communication and decision making during the pandemic and after.

Telehealth has greatly expanded the abilities of patients to see clinicians remotely or for clinician to clinician consultation, but prior to COVID-19 there were few interventions aimed at the family members of hospitalized patients. We feel we are poised to rapidly move along the NIH research pathway given that we are studying our early implementation. At the conclusion of this pilot, we will then conduct an effectiveness trial, followed by an embedded, pragmatic clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* 65 years or older
* cognitive impairment due to ADRD, delirium, or other causes of cognitive impairment severe enough that they require a surrogate for all medical decisions
* must have a surrogate decision maker based on a previously executed healthcare representative form or based on Indiana statute.

Surrogate:

* English-speaking
* Surrogate does not plan to be at patient's bedside every day
* surrogate is 18 or older

Exclusion Criteria:

Patient:

* Less than 65 years old
* Incarcerated individuals (e.g. prisoners)
* Lack of cognitive impairment
* Terminal wean/ actively dying

Surrogate:

* Less than 18 years old
* Incarcerated individuals (e.g. prisoners)
* non-English speaking
* plans to be at patient's bedside every day
* has a care contract or flagged for security risk
* state-appointed guardians

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Measure change in ratings of communication quality among study participants using the FICS at baseline, 6-8 weeks after patient discharge, and 6 months after patient discharge | 6-8 weeks after discharge, 6 months after discharge
  Communication quality will be measured using the validated Family Inpatient Communication Survey (30 item scale)

SECONDARY OUTCOMES:
Measure change in participant depression among study participants using the PHQ-8 at baseline, 6-8 weeks after discharge, and 6 months after discharge | Baseline, 6-8 weeks after discharge, 6 months after discharge
  Depression will be measured using the validated Patient Health Questionnaire (8 item)
Measure change in anxiety among study participants using the GAD-7 at baseline, 6-8 weeks after discharge, and 6 months after discharge | Baseline, 6-8 weeks after discharge, 6 months after discharge
  Anxiety will be measured using the validated Generalized Anxiety Disorder-7
Measure change in the impact of events among study participants using the IES-R at 6-8 weeks after discharge and 6 months after discharge | 6-8 weeks after discharge, 6 months after discharge
  Impact of Events will be measured using the validated Impact of Events Scale
Measure complicated grief for study participants of patients who died at 6 months after discharge | 6 months after death
  Complicated grief will be measured using the validated Inventory of Complicated Grief
Measure change in participants' ratings of communication quality over time for the duration of the patient's hospital stay | Communication quality will be measured daily during the first week and twice a week thereafter for the duration of the hospital stay, up to 1 year
  Communication quality will be measured from participants responses to texted survey questions (ecological momentary assessment) written by the study team. Participants will respond on a 5 point Likert scale.

OTHER OUTCOMES:
Measure the change in observable and/or reported level of pain in patients of participants in the intervention group. | Pre/post observations of pain will occur at the time of study intervention, typically within 1 hour.
  Clinical measures will be obtained through direct observation of the patient by study nurses using the PAINAD scale or through patient self-report using the FACES Pain Scale
Measure the change in observable and/or reported level of distress in patients in the intervention group before and after study intervention | Pre/post observations of distress will occur at the time of study intervention, typically within 1 hour of each other.
  Clinical measures will be obtained by study nurses using the distress thermometer for patients who are able to self-report.
Measure the change in blood pressure in patients in the intervention group before and after study intervention | Pre/post observations of blood pressure will occur at the time of study intervention, typically within 1 hour of each other.
  The nurse will obtain the patient's blood pressure before and after the intervention
Measure the change in heart rate in patients in the intervention group before and after study intervention | Pre/post observations of heart rate will occur at the time of study intervention, typically within 1 hour of each other.
  The nurse will obtain the patient's heart rate before and after the intervention
Measure the change in respiratory rate in patients in the intervention group before and after study intervention | Pre/post observations of respiratory rate will occur at the time of study intervention, typically within 1 hour of each other.
  The nurse will obtain the patient's respiratory rate before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alexia M Torke, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No